CLINICAL TRIAL: NCT06850129
Title: Efficacy of a Digital Educational Intervention in Patients With Type 2 Diabe-tes Mellitus. A Multicenter, Randomized and Prospective 6-month Follow-up Study
Brief Title: Efficacy of a Digital Educational Intervention in Patients With Type 2 Diabetes Mellitus
Acronym: DDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HOSPITAL VITHAS SEVILLA (Network)
Responsible Party: Principal Investigator, Irene Caballero Mateos, PRINCIPAL INVESTIGATOR, HOSPITAL VITHAS SEVILLA
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: DIGITAL DIABETES COACH_V_1.0.0; acf93301039dc0d0207316e1a95891 (Other: FISEVI)
Record Dates: First submitted 2025-01-16; First posted 2025-02-27 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2025-02

CONDITIONS: Diabetes Mellitus Type 2
Keywords: tyoe 2 Diabetes Mellitus; digital; metabolic control; social networks
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: randomization was carried out by a person external to the study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Non intervention, usual parctice (No Intervention): Usual practice
- digital intervention (Experimental): Behavioral: diabetes eduaction This was a multicenter, randomized, prospective study that included adults with type 2 diabetes with poor metabolic control, who started treatment with GLP-1 receptor agonists, with the ability to use digital tools, especially via smartphone. Patients were randomly assigned to either a digital intervention group or a usual care group. The intervention group received education through social networks and digital tools (pedometer activation, sending healthy habits guide-lines), in a structured program of healthy lifestyle changes. All this, through the figure of a "Digital Coach" for weekly and on-demand advice and support on an individualized basis. Baseline and follow-up data were collected on demo-graphic characteristics, clinical parameters, treatment adherence, and quality of life.
  Interventions: Behavioral: DIGITAL INTERVENTION

INTERVENTIONS:
Behavioral: DIGITAL INTERVENTION — All patients received specific information about DM, treatments and po-tential complications. Then, patients were randomized to the digital interven-tion group or usual care. Those patients randomized to the intervention group were educated in the use of different social networks with access to infor-mation related to healthy lifestyle habits, dietary support, optimization of physi-cal activity, insulin titration, therapeutic targets, self-care, based on validated material from scientific societies and endorsed in diabetes education. Patients also had the valuable resource of a Digital Diabetes Coach: an online expert specializing in therapeutic education. This virtual guide provided patients with the flexibility to interact in both unidirectional and bidirectional ways, using methods such as chat boxes, audio messages, videos, and more. Through this digital medium, patients could seek guidance and have their questions re-solved.
  Other Names: DIDITAL DIABETES COACH
  Arms: digital intervention

SUMMARY:
The goal of this interventional study is to evaluate the change in the HbA1c value, changes in body composition and evaluation of response using validated questionnaires of satisfaction with healthcare professionals during 6 months follow-up.

The primary purpose of the study is to observe whether patients with a poor control of Diabetes type 2, in the digital intervention group through social networks can improve the control of their disease with quantifiable analytical values, as well as enhance their knowledge of the disease and its treatment, achieve greater satisfaction with healthcare professional and improve adherence to treatment.

The primary hyphotesis is that people with Type 2 Diabetes who participate in an educational intervention through digitalized systems and social networks achieve better metabolic control, including a reduction in HbA1c levels, improve their quality of life, expand their knowledge about disease management, and reduce healthcare resource utilization.

DETAILED DESCRIPTION:
This was a multicenter, randomized, prospective and interventional study that included adults with T2DM that started treatment with GLP-1 receptor agonists, had poor metabolic control (HbA1c >7%), were able to use a smartphone-based home digital tool, and access to social networks and webinars focus on diabetes education. In addition, the patients had to be on stable doses of oral antidiabetics for at least the previous 90 days. By contrast, patients with lack of motivation or unable to use social networks, unable to read or write in Spanish, previous history of psychiatric disorder or serious organic disease, using systemic corticosteroids (>10 days in treatment), or being pregnant, were excluded. Outpatients were recruited during one year from the Endocrinology Depart-ments of the Virgen Macarena Hospital (Seville), and Juan Ramón Jiménez Hospital (Huelva).

All patients received specific information about DM, treatments and potential complications. Then, patients were randomized to the digital intervention group or usual care. Those patients randomized to the intervention group were educated in the use of different social networks with access to information re-lated to healthy lifestyle habits, dietary support, optimization of physical activity, insulin titration, therapeutic targets, self-care, based on validated material from scientific societies and endorsed in diabetes education. Patients also had the valuable resource of a Digital Diabetes Coach: an online expert specializing in therapeutic education. This virtual guide provided patients with the flexibility to interact in both unidirectional and bidirectional ways, using methods such as chat boxes, audio messages, videos, and more. Through this digital medium, patients could seek guidance and have their questions resolved. The Digital Diabetes Coach operated under the supervision of a multidisciplinary team, endocrinologists, nutritionists, and certified diabetes educators. This team en-sured that patients received comprehensive support and guidance tailored to their individual needs. Patient interactions were facilitated through a variety of digital platforms, which were selected based on the patient's preferences and in consultation with their Digital Diabetes Coach. These interactions aimed to provide essential support and motivation for patients. The communication channels employed included email, Skype, WhatsApp, telephone calls, and video conferencing, allowing for flexibility and convenience in connecting with patients. The main communication channels used in this study included tele-phone calls, WhatsApp, email and Skype video calls. Among them, WhatsApp was the preferred application by patients to ask questions and share information with professionals, regardless of their educational and socioeconomic level. Patients with higher educational levels also felt comfortable with communication through videoconferencing, while this medium was not the most desired by patients with a lower educational level or those from rural areas. In addition, webinars through Instagram in real time or recorded were also used. Furthermore, a comprehensive diabetes education program was introduced on a weekly basis, with 30-45 minutes sessions. This program covered a wide spectrum of critical topics, including proper injection techniques, dosage adjustments for medications, strategies for managing adverse events, personalized recommendations for physical activity, guidance on blood glucose profiling and interpretation, strategies for handling hypoglycemia and hyperglycemia, portion controlled dietary plans, and insights into potential health conditions associated with poor macro and microvascular control. The educational materials used for these sessions were sourced from scientific societies, external companies endorsed by these societies, as well as materials developed by our center. To ensure effective communication and timely assistance, a two-way communication system was established. Patients were encouraged to seek answers to their questions and access information on-demand through messenger apps and other digital platforms. This approach allowed for a responsive and patient-centered approach to addressing individual needs and concerns. During the different interventions, patients were promoted to send data on weight, capillary blood glucose, activation of pedometers on their mobile phone etc.

In the control group, visits to the specialists (i.e., endocrinologist) were performed every 3 months, that included diabetes education intervention by the nursing staff (i.e., use of medication, adherence to treatment and basic guidelines for the management of their diabetes), for around 30 minutes in each consultation.

At baseline, demographic data, educational level, employment status, physical examination, treatment for diabetes (total insulin dose), and analytical data within the 12 weeks before inclusion were collected. Data was obtained from each electronic clinical history and glucose levels from the Libreview system. During the intermediate visit (3 months±15 days from base-line), physical examination, number of scans, adherence, verification that the patient adequately understood the material delivered and made use of social networks, changes of treatment, regular diabetes education, and adverse events since last visit were recorded. As this was a routine visit, the education activities by the staff (nursing and endocrine specialist) were homogeneous in both groups. At study end (6 months±15 days from baseline), physical examination, number of scans, adherence, verification that the patient adequately understood the material delivered and made use of social networks, changes of treatment, regular diabetes education and adverse events since last visit were recorded. For changes of treatment, the total dose of insulin was considered, rather than maximum or minimum doses of insulin. Changes in body composition along the study were also analyzed, including body fat mass, visceral fat area, fat-free mass and skeletal muscle mass, through segmental analysis of multi-frequency bioelectrical impedance (SMF-BIA; Inbody 770, In-body Co,Ltd, Korea).

Additionally, at baseline and at study end, different validated questionnaires were fulfilled by the patients.

The Quality of Life was evaluated with the Spanish version of the Diabetes Quality of Life Questionnaire (EsDQOL). This questionnaire has 4 sections: satisfaction (15 questions, with a score that ranges from 1 [very satisfied] to 5 [not at all satisfied]; 15 points implies great satisfaction), im-pact (17 questions, with a score that ranges from 1 [never] to 5 [always]; 17 points indicates that DM has little impact on daily life), social/vocational concerns (7 questions, with a score that ranges from 1 [never] to 5 [always]; 7 points indicates that DM causes little worry on a daily basis), and DM re-lated concerns (4 questions, with a score that ranges from 1 [never] to 5 [al-ways]; 4 points indicates that diabetes causes little worry on a daily basis).

The knowledge that DM patients had of diabetes was evaluated by the ECODI scale (scale of knowledge about diabetics). This scale has 25 items with 4 possible answers.

The eight items of Clarke's questionnaire were used to evaluate the perception about hypoglycemia. This scale has a total score of 0 to 7. Higher scores indicate diminished awareness.

The 4-item Morisky-Green scale was used to evaluate medication adherence. This scale has a total score of 0 to 4. A score of four denotes high adherence.

Patient's healthcare experience was assessed with the "Instrument for Evaluation of the Experience of Chronic Patients" (IEXPAC) questionnaire. This is a self-administered, 12-item, multiple-choice questionnaire. Items 1 to 10 describe the patient's experience in the last six months in three domains (productive interactions, new model of the patient's relationship/interaction with the healthcare system, and patient's self-care). The last 2 questions only apply to patients who have been hospitalized, not be-ing counted in the total of answers. As a result, the overall score ranges from 0 (worst experience) to 10 (best experience).

ELIGIBILITY:
Inclusion Criteria:

* Adults with T2DM that started treatment with GLP-1 receptor agonists (more tha 18 years)
* Poor metabolic control (HbA1c >7%)
* Were able to use a smartphone-based home digital tool, and access to social networks and webinars focus on diabetes education.
* Stable doses of oral antidiabetics for at least the previous 90 days before the have signed the Inform consent form.

Exclusion Criteria:

* Patients with lack of motivation or unable to use social networks
* Unable to read or write in Spanish
* Previous history of psychiatric disorder or serious organic disease
* Using systemic corticosteroids (>10 days in treatment)
* Being pregnant or possibility to be during the clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2020-10-26 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2023-10-26 (Actual)

PRIMARY OUTCOMES:
weight in Kilograms | From enrollment to the end of treatment at 6 months
  Participants' weight will be measured in a fasting state, with an empty bladder, and wearing light clothing. The measurement will be conducted using calibrated devices to ensure accuracy.
Hba1c in percent (lab result) | From enrollment to the end of treatment at 6 months
  HbA1c levels will be measured through blood analysis to assess the degree of long-term glycemic control in patients
weight and height will be combined to report BMI (Kg/m^2) | From enrollment to the end of treatment at 6 months
  his measurement will provide an assessment of the participant's body composition

SECONDARY OUTCOMES:
FPG (Fasting plasma glucose) in mg/dl | From enrollment to the end of treatment at 6 months
  lab results
total insulin in UI (international units) | From enrollment to the end of treatment at 6 months
  lab results

CONTACTS AND LOCATIONS:
Overall Officials: Angel Vilches Arenas, Phd, Study Director — Fundación Pública Andaluza para la gestión de la Investigación en Sevilla
Locations (2):
- Spain (2):
  - Hospital Vithas Sevilla, Seville, Castilleja de LA Cuesta
  - Fundacion Vithas, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Caballero Mateos I, Morales Portillo C, Lainez Lopez M, Vilches-Arenas A. Efficacy of a Digital Educational Intervention for Patients With Type 2 Diabetes Mellitus: Multicenter, Randomized, Prospective, 6-Month Follow-Up Study. J Med Internet Res. 2025 Apr 10;27:e60758. doi: 10.2196/60758. PMID 40209213